CLINICAL TRIAL: NCT03815526
Title: The Immediate Effects of Applying Dynamic Tape, Kinesio Tape and Sport Tape With Chronic Ankle Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: N201811015
Record Dates: First submitted 2019-01-09; First posted 2019-01-24 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-01

CONDITIONS: Taping; Ankle Sprains
Keywords: DynamicTape; Sport Tape; Kinesio Tape
MeSH Terms: conditions — Ankle Injuries | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dynamic tape (Experimental)
  Interventions: Other: Dynamic tape
- Kinesio tape (Experimental)
  Interventions: Other: Kinesio tape
- Sport tape (Experimental)
  Interventions: Other: Sport tape

INTERVENTIONS:
Other: Dynamic tape — Dynamic tape apply 1 time
  Arms: Dynamic tape
Other: Kinesio tape — Dynamic tape apply 1 time
  Arms: Kinesio tape
Other: Sport tape — Dynamic tape apply 1 time
  Arms: Sport tape

SUMMARY:
Injuries to the ankle joint account for 20% of the population that is afﬂicted with joint injury and the largest percentage of self-reported musculoskeletal injuries (> 10%) are to the ankle. Ankle sprain has a large portion in ankle injuries and occurs not only in the sporting population but also in the general community. Although the acute symptom would be resolve quickly, but many people still report persisting problems, such as pain and instability. Chronic ankle instability (CAI) is one of the most common of these residual problems.

Kinesio Tape and White Duck Tape are often applied in patients with CAI, attempt to increase the ankle joint stability, and improve motor performance. However, the previous studies had controversial result to the effects of kinesio tape and white duck tape. The previous studies also showed the insufficient of supporting force and elasticity of kinesio tape and white duct tape. The Dynamic Tape was developed by Kendrick in 2009, which refined the characteristic of elasticity and supporting force.

Therefore the purpose of study is to comparison the effects of static and dynamic balance performance, weight shifting ability and functional movement between kinesio tape, white duck tape and dynamic tape when applied on patients with CAI. With the result may provide an optical method to increase the movement performance of patients with CAI.

The study suspected to recruit 90 volunteers with CAI, and randomly divided to three different groups: Kinesio tape group, White duck tape group and Dynamic tape group. We make postural stability test and limit postural stability test with Biodex Balance System (SD), Y-balance test and single leg hop test to both affected side and sound side foot before applying the tape. After applying the tape according to the divided group, we will repeat the test above again. We will compare the results of the test between groups and within groups.

ELIGIBILITY:
Inclusion Criteria:

1. A history of at least one signiﬁcant ankle sprain

   * The initial sprain must have occurred at least 12 months prior to the study enrolment
   * Was associated with inﬂammatory symptoms (pain, swelling, etc)
   * Created at least one interrupted day of desired physical activity
2. A history of the previously injured ankle joint 'giving way' , and /or recurrent sprain and/or 'feelings of instability'.

Exclusion Criteria:

1. A history of previous surgeries to the musculoskeletal structures (ie, bones, joint structures and nerves) in either lower extremity.
2. A history of a fracture in either lower extremity requiring realignment.
3. Acute injury to the musculoskeletal structures of other joints of the lower extremity in the previous 1 months, which impacted joint integrity and function (ie, sprains, fractures) resulting in at least 1 interrupted day of desired physical activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Biodex Balance System | 1 day
  Overall Stability Index, Anterior/Posterior Index, Medial/Lateral Index Limits of stability direction control score (Overall, Forward, Backward, Right, Left, Forward/Right, Forward/Left, Backward/Right, Backward/Left)

SECONDARY OUTCOMES:
Y-balance test | 1 day
  dynamic reach (cm): anterior, posterior/medial, posterior/lateral
Single leg hop test | 1 day
  single leg hop laterally distance (cm) and 15 cm side hop time(second)

CONTACTS AND LOCATIONS:
Locations (1):
- Wanfang Hospital, Taipei, Taiwan